CLINICAL TRIAL: NCT03663894
Title: Clinical Characteristics and Outcomes of Relapsed Follicular Lymphoma After Autologous Stem Cell Transplantation at Rituximab Era
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: ASCT Sesques
Record Dates: First submitted 2018-08-22; First posted 2018-09-10 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Patient's Outcome Prognostic Factors
Keywords: Autologous stem cell transplantation; rituximab; Follicular Lymphoma; prognosis
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Introduction High dose chemotherapy followed by Autologous Stem Cell Transplantation (ASCT) is a therapeutic option in follicular Lymphoma after first line treatment failure. The clinical characteristics and outcome of FL patients who relapsed after HDT+ASCT and therapeutic management in the rituximab era are not well known and may represent a difficult challenge.

Patients and Methods: The investigators conducted a retrospective analysis of FL patients who relapsed after HDT+ASCT in four French centers treated between 2000 and 2014. Clinical records were reviewed for clinical characteristics and treatment strategy at relapse. The investigators aimed to identify prognostic factors related to patient's outcome.

ELIGIBILITY:
Inclusion Criteria:

* they were older than 18 years
* presented FL at diagnosis (Grade 1, 2, or 3a).
* received high-dose therapy (HDT) with ASCT from 2000 to 2014

Exclusion Criteria:

1. they had already been treated with a 1st ASCT,
2. had a previous history of histological transformation before ASCT
3. if they were rituximab naive prior to ASCT.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 95 consecutive patients who fulfilled the eligibility criteria for this study were reviewed retrospectively with data cut-off of December 2014. FL patients in relapse after ASCT. All patients presented at diagnosis a grade 1, 2, or 3A follicular lymphoma confirmed by either excisional or core needle biopsy.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2017-07-30 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Survival after relapse (SAR) post ASCT in follicular lymphoma | Year 6
  Factors that predicted SAR

SECONDARY OUTCOMES:
Histological Transformation at relapse | Year 6
  A biopsy was performed at the first relapse or progression after ASCT.
treatment of relapse | Year 6
  Chemotherapy, radiotherapy…

CONTACTS AND LOCATIONS:
Overall Officials: Pierre SESQUES, MD, Study Director — Hospices Civils de Lyon
Locations (1):
- Centre Hospitalier Lyon Sud, Hematology department, Pierre-Bénite, France